CLINICAL TRIAL: NCT07044752
Title: Paterson Prevention Project Anxiety Prevention Intervention
Brief Title: Step 1: Be Aware, Anxiety Prevention Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000030293
Record Dates: First submitted 2025-06-03; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Moderate Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anxiety Intervention (Other): 5-educational session anxiety intervention for teens
  Interventions: Behavioral: Anxiety Prevention Intervention; Behavioral: Anxiety Intervention

INTERVENTIONS:
Behavioral: Anxiety Prevention Intervention — community and school based, delivered by peers from the community to educate and lower anxiety symptoms among youth
Behavioral: Anxiety Intervention — 5-session social and behavioral intervention about managing anxiety symptoms

SUMMARY:
Youth of color, particularly in urban communities, face disproportionate anxiety levels due to systemic inequities, including exposure to violence, economic instability, and neighborhood disadvantage. Despite increased need, these communities often lack accessible, culturally relevant mental health interventions. This study presents a protocol for a community-driven anxiety prevention intervention tailored to urban youth of color using community-based participatory research (CBPR) methods. The intervention, co-developed with community partners and youth includes five structured weekly sessions on psychoeducation, coping skills, and role-playing exercises. Facilitators trained in social work or psychology will deliver the intervention, with at least one facilitator from the target community ensuring cultural relevance. Recruitment will occur through collaboration with a local high school, with counselors identifying high-risk youth. Data from pilot interventional trial will be collected at baseline, post-intervention, and a three-month follow-up using validated measures such as the Generalized Anxiety Disorder-7 (GAD-7) scale. This study highlights community-based participatory research approach in addressing mental health disparities among urban youth. By incorporating community perspectives, the intervention ensures cultural alignment. Findings will inform future adaptations of community centered anxiety interventions and contribute to knowledge on improving mental health accessibility for marginalized youth. If effective, this model could be expanded to support youth in other under-resourced communities.

ELIGIBILITY:
Inclusion Criteria:

* able to speak and read in English
* reside in Paterson

Exclusion Criteria:

* English is not first language and cannot read or write English
* Does not have residence in Paterson
* Has not provided consent to participate in study

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder | 30 days
  Symptoms of Anxiety, Mild, Moderate, Severe

CONTACTS AND LOCATIONS:
Overall Officials: Ijeoma Opara, PhD, Principal Investigator — Yale University
Locations (1):
- Paterson College Achieve High School, Paterson, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No